CLINICAL TRIAL: NCT05387408
Title: Improving Health and Employment Outcomes Through Workplace Opioid Policies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201912063
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid Use Disorder; Construction Industry
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participating union health fund (Other): The investigators will recruit three health funds into a single arm trial. Each health fund will receive the intervention, "Workplace Opioid Prevention Guidelines." The intervention is a set of guidelines containing information and suggested changes the health fund may make to their health and safety program specifically to prevent and manage opioid abuse in their workforce. The health fund the investigators receive the intervention after completing baseline data collection. The investigators will provide assistance with using the intervention as needed over a 6 month period of time, and measure changes the health fund makes to their health and safety program based on information in the guidelines. At 6 months, the investigators will repeat baseline data collection for the efficacy trial.
  Interventions: Behavioral: Best Practice Health and Employment Opioid-related Policies

INTERVENTIONS:
Behavioral: Best Practice Health and Employment Opioid-related Policies — The intervention will include information to promote policies and programs to prevent opioid abuse and aid recovery such as drug testing for opioids, health and employee assistance programs, job accommodations, and education to deliver training to prevent opioid use, and prevent stigma.

SUMMARY:
Evaluate the feasibility of implementing workplace opioid guidelines in the construction trades; define and collect measures of implementation and efficacy. The investigators will implement the intervention in three local union health funds, evaluate the implementation using the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework, and collect the data needed to measure the efficacy of health changes due to implementation of the intervention (workplace opioid guidelines). This is only a feasibility trial in preparation for conducting an randomized control trial. For the efficacy trial, the investigators will measure pre-post health change using two data sources: 1) administrative health claims and electronic member work hours, and 2) worker/member surveys. To monitor implementation of the intervention, the investigators will measure changes made to the health funds opioid prevention program through qualitative interviews with the health fund manager and through worker surveys for worker awareness and use of the health fund program changes pre-post implementation. The efficacy outcomes for the administrative health (and pharmacy) claims and work hours record will measure opioid prescriptions, chronic opioid use, and OUD in health claims and pharmacy data (details below). The efficacy outcomes for the worker surveys will record changes in misuse of opioids, change in missed days/work productivity, change in attitudes toward seeking help if worker was struggling with opioid misuse, and awareness and use of health fund programs (i.e. employee assistance programs, healthcare recovery services). the investigators will collect data at baseline and and after 6 months for the study of implementation and efficacy (a pre/post design, one-arm trial).

DETAILED DESCRIPTION:
We will recruit three health funds to implement the opioid guidelines. Participating health funds will receive an introduction to the intervention materials and will discuss guideline adoption procedures with the research team. In order to implement the workplace opioid guidelines (intervention), each participating health fund must agree to make changes to their health fund policies and to engage employers to change some of the workplace policies. In order to evaluate the guideline implementation, the health funds must participate in baseline, 6, and 12 month interviews to describe changes in their opioid policies and programs, distribute a survey link to their members, and provide access to their health claims, pharmacy data, and employee work hour records. Participating health funds will be asked to sign a partnership agreement form, as we have done in our past intervention studies with construction partners, to show their understanding of the project and their agreement to participate in all study activities and to provide data over the course of the implementation trial.

We will use the RE-AIM framework to assess the Reach, Adoption, Implementation, and Maintenance of the intervention in each participating health fund. Reach will assess workers' awareness of policies and benefits, Adoption will identify the new policies agreed to by the board of trustees for each health fund, Implementation will describe the strategies for enacting the adopted policies and programs, and the extent these strategies are implemented, and Maintenance will identify the continued delivery of implemented policies and programs. Adoption, Implementation, and Maintenance will be assessed via periodic interviews with the health fund partners. Collection of health fund data on claims and work hours will show the feasibility of obtaining and using these data to evaluate effectiveness in the planned future study. Use of the RE-AIM framework will provide an evaluation of the extent to which the opioid guidelines are implemented, and describe barriers to implementation.

Data collection for the outcome measures will include worker surveys and health claims from the enrolled union health funds. We will analyze the data by measuring the pre-post change in the outcome measures. Participating health funds will provide access to construction workers to collect a cross-sectional sample of surveys at three points in time. We will ask our partners to distribute a link for a Redcap survey to a representative sample of their members (eligible workers) with a goal of at least 300 returned surveys per health fund at baseline. We will collect an additional 300 surveys at 6 months (and at 12 months if time allows) from each fund after initiating the intervention. We will attempt to oversample women and minorities, as they are less common in this worker population. The brief survey will ask about workers' knowledge of their health fund's benefits and policies, attitudes toward use of opioids by self and others, employment status, participation in union programs including EAP, and health-related productivity using widely used survey instruments. We will work with participating funds to obtain health claims and pharmacy data for all eligible union members for a period of at least 3 years prior to implementation of the intervention. From health claims, we will request data for demographics, dates of service, and diagnoses and procedure codes. From pharmacy data we will request the dates of prescription fill, drug name, days' supply, and fill quantity. From merged claims and pharmacy data we will identify relevant opioid use case definitions: workers who received opioid prescriptions, workers who misused opioids (defined as multiple prescriptions of opioids in a single visit, overlapping supply of opioids, early refills), workers who received chronic opioid prescriptions (classified as 60 day supply in a 90 day period), and workers with OUD (defined as a diagnostic code of F11, poisoning T40, or prescription for MAT). We will also work with the funds to obtain employee work hour records. Using the same unique identifier as the health claims data, we will link claims and pharmacy data to the weekly or monthly work hour logs, union eligibility status (active/retired/other), and employer. We will examine loss of employment or average work hours for those who remain employed among workers who meet or do not meet one of the opioid use case definitions. We will collect other administrative data including the number of visits to the employee assistance program (EAP), the number of workers who enrolled in recovery centers, and those filing for disability benefits to compare utilization of services by workers before and after the intervention.

We will measure the change from baseline (pre-) to 6 months (post-) and 12 months (post- if time allows). The outcome measures will be from claims data (pre-post change in opioid misuse, chronic opioid use, and opioid use disorders) and from surveys (opioid misuse, lost time due to pain, and worker willingness to seek help). For claims data, we will compare the prevalence of the outcomes from 3-year period prior to the intervention compared to the 6-months after start of the intervention (collected at 6-months). For survey data, we will compare the prevalence of the outcomes from cross-sectional data collected at baseline to cross-sectional data collected at 6-months after start of the intervention. We will collect surveys from 300 members of the population, representative of the characteristics of the population, at baseline and at 6-months (and 12months if time allows).

To learn about changes each participating health fund makes to their health and safety program from using the Opioid Guidelines, we will interview the health administrator at baseline, before starting the intervention, will meet monthly with the administrator to learn about changes to their program, and conduct a final assessment. We will explore what plans the health fund wants to make to reduce opioid abuse among their members, the steps they take toward implementing changes including their strategies and response to their actions. We will also document the barriers encountered while trying to make plans and take action for change.

ELIGIBILITY:
Inclusion Criteria:

* members enrolled in union health funds

Exclusion Criteria:

* none.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4939 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Dale, Ph.D, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to make the data from the worker surveys available to other researchers. The available data fill be de-identified surveys of a representative sample of union members from health funds collected at two time points on (1) pain and opioid use (2) missed days related to health and opioid use, (3) workers' knowledge of their health fund's benefits and policies, (4) self-reported use of benefits, and (5) attitudes toward use of opioids by self and others. This data will be made publicly available through the Helping to End Addiction Long-Term (HEAL) Initiative Central Data Repository. The investigators will work with the repository to prepare the data and accompanying instructions. The investigators have submitted the data for review as of 11/10/23.
Supporting Information: ICF, Analytic Code
Time Frame: The data is under review at the data sharing center as of 11/10/23. We anticipate the data will be available by March 2024. There is no expiration date.
Access Criteria: The de-identified data has been shared with the Interuniversity Consortium for Political and Social Research (ICPSR) group at the University of Michigan. There is no restrictions from the research team at Washington University. Any access criteria would be at the discretion of the ICPSR group.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We started recruiting health funds in February 2022, with 3 health funds seeking to participate by May 2022. Health Fund A enrolled at the end of May 2022, health fund B enrolled at the end of July, but health fund C never completed the enrollment so was dropped in November 2022.
Groups:
- Single Arm/ Participating Union Health Funds: Enrolled health funds were to provide administrative claims (deidentified medical and pharmacy claims with a linking variable) at baseline for primary outcome. They were to invite a representative group of their members to complete the worker survey (to collect 300 surveys/health fund). Follow up data for administrative claims for 6-months and worker surveys at 6 months were to be collected after a 6-month trial of the intervention. The intervention trial was for the health fund administrator to use the Workplace Guidelines to Prevent Opioid Abuse in the Construction Trades, created as part of this R34 study and to be part of the feasibility trial for this study.
Period: Overall Study
Arm/Group | Single Arm/ Participating Union Health Funds
Started | 4939 (Health fund A had 4881 members in the administrative claims data (of whom 69 members completed the worker survey). Health fund B did not provide claims data but had 58 members complete the worker survey.)
Completed | 0 (There was no follow up data collected for this study as Health Fund A did not have time to provide administrative claims after 1 year and collection of surveys was not successful enough at baseline to warrant a second data collection. Health Fund B did not provide the researchers with their administrative data, and their low participation of members completing the baseline survey did not warrant a second data collection.)
Not Completed | 4939
Not completed — Lack of time and access to participants to complete the survey by the health fund administrators | 4939

BASELINE CHARACTERISTICS:
Population: The participants came from 2 health funds: from health fund A, there were 4881 members (4881 in the administrative dataset, and 69 from worker surveys); from health fund B, there were 58 members, (n=58 from worker surveys). The third health fund did not complete enrollment into the study.
Arm/Group | Participating Union Health Fund
Number analyzed (Participants) | 4939
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The data came from two health funds and includes claims/surveys from Fund A and surveys from Fund B.
  years | 42.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: four participants did not complete the item on gender.
  Participants
    number analyzed (Participants) | 4935
    Female | 265
    Male | 4670
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The health claims data from the health fund A did not collect race, however we did request race for the worker surveys from the health fund A. There were 69 worker surveys completed from health fund A, and 58 surveys completed from health fund B for a total of 127 surveys. We are presenting the race information from only the survey data.
  Participants
    number analyzed (Participants) | 127
    American Indian or Alaska Native | 1
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 6
    White | 111
    More than one race | 1
    Unknown or Not Reported | 8
Opioid misuse by claims data [Count of Participants; unit: Participants] — After combining the medical and pharmacy claims, each "treatment" was determined by the diagnosis code and date of service. Opioid prescriptions were linked to treatments. Opioid misuse was defined by an overlap in opioid prescription fills (early refills) or multiple fills on the same day by different providers. Chronic use was defined by receiving more than 60 days supply of medications in a 90 day window. Opioid use disorder was defined by an ICD-10 T40 (Poisoning) &/or F11 (opioid related disorders) &/or prescribed medication assisted treatment including "methadone" or "buprenorphine". Population: Claims data only came from health fund A.
  Participants
    Opioid misuse: number analyzed (Participants) | 4881
    Opioid misuse | 209
    Chronic opioid use: number analyzed (Participants) | 4881
    Chronic opioid use | 121
    Opioid use disorder: number analyzed (Participants) | 4881
    Opioid use disorder | 85
Opioid misuse by worker surveys [Count of Participants; unit: Participants] — The survey contained items that were used to define opioid misuse if a member responded yes to one of the following items: took more opioids than prescribed, took opioids longer than prescribed, took opioids prescribed to someone else, or for a reason other than pain relief. Population: Each health fund shared communication and the survey link throughout their membership, through repeated communications in one or more methods (email, newsletter, word of mouth). At baseline, we collected 69 surveys from health fund A and 58 surveys from health fund B.
  Participants
    number analyzed (Participants) | 127
    (all) | 23
Lost time due to pain on worker survey [Count of Participants; unit: Participants] — The worker surveys were sent out to two health fund via a survey link or QR code. The survey contained one item asking the member if they had "missed workdays due to pain". Population: Each health fund shared communication and the survey link throughout their membership, through repeated communications in one or more methods (email, newsletter, word of mouth). At baseline, we collected 69 surveys from health fund A and 58 surveys from health fund B.
  Participants
    number analyzed (Participants) | 127
    (all) | 22
Worker willingness to seek help if struggling with opioids [Count of Participants; unit: Participants] — The worker survey will assess whether the member perceives that if the person was struggling with opioid misuse or a substance use problem, the member would be willing to seek help through 1) their workplace (seek help from a supervisor, someone from human resources, ask a trusted coworker for help, attend an alcoholics or narcotics anonymous group or meet with a peer specialist), or 2) professional help including an employee assistance program or behavioral health. Population: Each health fund shared communication and the survey link throughout their membership, through repeated communications in one or more methods (email, newsletter, word of mouth). We collected 69 surveys from health fund A and 58 surveys from health fund B.
  Participants
    number analyzed (Participants) | 127
    (all) | 98

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Workers With Opioid Misuse, Opioid Use Disorder and Opioid Overdose: Administrative Data [Primary Outcome]
Description: Problem opioid use is a composite outcome of opioid misuse, OUD, or opioid overdose. The investigators will use health and pharmacy claims data to identify workers who misused opioids (defined as multiple prescriptions of opioids in a single visit, overlapping supply of opioids, early refills), workers who received chronic opioid prescriptions (classified as 60 day supply in a 90 day period), and workers with Opioid Use Disorder (OUD) (defined as a diagnostic code for OUD or opioid overdose (ICD10=F11 or T40), or a prescription for Medication Assisted Treatment such as buprenorphine, naltrexone or methadone).
Time Frame: The investigators will collect administrative data to assess change over time (change of opioid misuse and OUD at 6 months following delivery of the intervention).
Population: We were unable to collect outcome data at 6 months so are unable to analyze change from baseline.
Groups:
- Single Arm/ Participating Union Health Funds: The investigators planned to recruit three health funds into a single arm trial. Each health fund will receive the intervention, "Workplace Opioid Prevention Guidelines." The intervention is a set of guidelines containing information and suggested changes the health fund may make to their health and safety program specifically to prevent and manage opioid abuse in their workforce. The health fund the investigators receive the intervention after completing baseline data collection. The investigators will provide assistance with using the intervention as needed over a 6 month period of time, and measure changes the health fund makes to their health and safety program based on information in the guidelines. At 6 months, the investigators will repeat baseline data collection for the efficacy trial (collecting the administrative claims and worker surveys at follow up).
  Best Practice Health and Employment Opioid-related Policies: The intervention will include information to promote policies and programs to prevent opioid abuse and aid recovery such as drug testing for opioids, health and employee assistance programs, job accommodations, and education to deliver training to prevent opioid use, and prevent stigma.
Arm/Group | Single Arm/ Participating Union Health Funds
Number analyzed (Participants) | 0

2. Primary Outcome: Proportion of Workers With Opioid Misuse: Worker Surveys
Description: The investigators will assess workers' misuse of prescription opioids (taking more than prescribed, longer than prescribed, prescribed to someone else or for a reason other than pain), (n=600 anticipated from 2 participating health funds)
Time Frame: The investigators will compare change at 6 months post-intervention (change of opioid misuse) of group-level data collected from groups of health fund members.
Population: Only two health funds participated, and each were unsuccessful to collect 300 surveys at baseline. The health funds did not attempt to collect 6 month survey data so no measure of change could be calculated.
Groups:
- Participating Union Health Funds: The investigators will recruit three health funds into a single arm trial. Each health fund will receive the intervention, "Workplace Opioid Prevention Guidelines." The intervention is a set of guidelines containing information and suggested changes the health fund may make to their health and safety program specifically to prevent and manage opioid abuse in their workforce. The health fund the investigators receive the intervention after completing baseline data collection. The investigators will provide assistance with using the intervention as needed over a 6 month period of time, and measure changes the health fund makes to their health and safety program based on information in the guidelines. At 6 months, the investigators will repeat baseline data collection for the efficacy trial.
  Best Practice Health and Employment Opioid-related Policies: The intervention will include information to promote policies and programs to prevent opioid abuse and aid recovery such as drug testing for opioids, health and employee assistance programs, job accommodations, and education to deliver training to prevent opioid use, and prevent stigma.
Arm/Group | Participating Union Health Funds
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Workers With Lost Time: Worker Surveys [Secondary Outcome]
Description: The investigators will assess workers' b) missed workdays due to pain/due to being high or recovering from night before, and (n=1800 anticipated)
Time Frame: The investigators will compare change at 6 months post-intervention (change in lost time) of group-level data collected from groups of health fund members.
Population: as for outcome 2
Arm/Group | Participating Union Health Fund
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Workers Who Are Willing to Seek Help: Worker Surveys [Secondary Outcome]
Description: The investigators will assess if workers' were struggling with opioid misuse/substance use problem, how willing the worker would be to seek help through 1) their workplace, 2) professional help (employee assistance program or behavioral health) (n=1800 anticipated)
Time Frame: The investigators will compare change at 6 months post-intervention (change of willingness to seek help) of group-level data collected from groups of health fund members.
Population: as for outcome 2
Arm/Group | Participating Union Health Funds
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Description: Primary data was collected through surveys but no identifiers were obtained. This study was considered minimal risk. The only way the researchers would learn about an adverse event is if the participating health fund shared this information.
Groups:
- Single Arm/ Participating Union Health Funds: The investigators will recruit three health funds into a single arm trial. Each health fund will receive the intervention, "Workplace Opioid Prevention Guidelines." The intervention is a set of guidelines containing information and suggested changes the health fund may make to their health and safety program specifically to prevent and manage opioid abuse in their workforce. The health fund the investigators receive the intervention after completing baseline data collection. The investigators will provide assistance with using the intervention as needed over a 6 month period of time, and measure changes the health fund makes to their health and safety program based on information in the guidelines. At 6 months, the investigators will repeat baseline data collection for the efficacy trial.
  Best Practice Health and Employment Opioid-related Policies: The intervention will include information to promote policies and programs to prevent opioid abuse and aid recovery such as drug testing for opioids, health and employee assistance programs, job accommodations, and education to deliver training to prevent opioid use, and prevent stigma.
Arm/Group | Single Arm/ Participating Union Health Funds
All-Cause Mortality (participants affected / at risk) | 0/4939
Serious Adverse Events (participants affected / at risk) | 0/4939
Other Adverse Events (participants affected / at risk) | 0/4939

LIMITATIONS AND CAVEATS:
Only two of the planned three health funds enrolled. Only one of the enrolled health funds provided administrative data but only for the 3-year period before the intervention (baseline). . Both of the enrolled health funds collected worker surveys at baseline but due to low participation, follow-up surveys were not collected. Only one of the health funds actively participated in implementing the intervention. High time demands, lack of access to data, and to members limited the study success.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT05387408/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT05387408/ICF_001.pdf